CLINICAL TRIAL: NCT01924260
Title: Phase I Study of the Combination of MLN8237 and Gemcitabine in Advanced Solid Tumors With Emphasis on Pancreatic Cancer
Brief Title: Alisertib and Gemcitabine Hydrochloride in Treating Patients With Solid Tumors or Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edward Kim (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Takeda (Industry)
Responsible Party: Sponsor-Investigator, Edward Kim, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 457403; UCDCC#240 (Other: UC Davis); P30CA093373 (NIH); X14020 (Other Grant/Funding Number: Takeda); NCI-2013-01388 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — MLN 8237; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (alisertib, gemcitabine) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and alisertib PO BID on days 1-3, 8-10, and 15-17. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alisertib; Drug: gemcitabine

INTERVENTIONS:
Drug: alisertib — Given PO
  Other Names: Aurora A kinase inhibitor MLN8237; MLN8237
Drug: gemcitabine — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; Gemzar

SUMMARY:
This phase I trial studies the side effects and the best dose of alisertib when given together with gemcitabine hydrochloride in treating patients with solid tumors or pancreatic cancer that is metastatic or cannot be removed by surgery. Alisertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving alisertib with gemcitabine hydrochloride may be an effective treatment for solid tumors or pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the feasibility and safety of MLN8237 (alisertib) when given in combination with gemcitabine (gemcitabine hydrochloride) to patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of MLN8237 when given in combination with gemcitabine to patients with advanced solid tumors and to recommend a phase II dose for the combination.

II. To obtain preliminary evidence of efficacy as judged by response rate and progression-free survival for this combination.

III. To investigate the pharmacokinetics of MLN8237 given in combination with gemcitabine in an expanded cohort of patients with pancreatic cancer.

OUTLINE: This is a dose-escalation study of alisertib.

Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1, 8, and 15 and alisertib orally (PO) twice daily (BID) on days 1-3, 8-10, and 15-17. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for dose escalation cohort: histologically or cytologically confirmed metastatic or unresectable solid tumor for which standard curative or palliative measures do not exist or are no longer effective
* Eligibility for the expansion cohort: histologically or cytologically confirmed metastatic or unresectable pancreatic adenocarcinoma for which curative treatment does not exist
* Zubrod (Eastern Cooperative Oncology Group [ECOG]) performance status 0 - 2
* Measurable or non-measurable disease. x-rays and/or scans for disease assessment of measurable disease must have been completed within 28 days prior to registration; non-measurable disease must also be assessed within 28 days prior to registration; (expansion - patients must have measurable disease)
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin within institutional normal limits
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 times institutional upper limit of normal or =< 5 times institutional upper limit of normal in the presence of liver metastases
* Creatinine =< 1.5 times institutional upper limit of normal OR

  * Creatinine Clearance >= 60ml/min/1.73m^2 measured by 24-hour urine collection
* Any number of prior chemotherapy regimens; up to two prior chemotherapy regimen in the palliative setting will be allowed in the expansion cohort. Prior gemcitabine-based regimes in the palliative setting are permitted if no evidence of progression on therapy or at least 6 months after discontinuation of gemcitabine based treatment. Prior gemcitabine in the adjuvant setting is permitted if last treatment was greater than 6 months prior to registration
* Any prior chemotherapy, immunotherapy or targeted therapy must have been completed at least 2 weeks prior to start of this protocol and all side effects (except alopecia, lymphopenia and hyperglycemia) resolved to grade 1 or less; any prior radiation must have been completed at least 2 weeks prior to start of therapy
* Pregnant or nursing women are ineligible; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document
* Ability to swallow and retain oral medications
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Male subject agrees to use an acceptable method for contraception during the entire study treatment period through 4 months after the last dose of MLN8237; male patients, even if surgically sterilized (ie, status postvasectomy) must agree to practice effective barrier contraception during the entire study treatment period and through four months after the last dose of study drug, or completely abstain from heterosexual intercourse

Exclusion Criteria:

* Prior treatment with Aurora A-targeted agents, including MLN8237
* History of Gilbert's syndrome
* Cardiac disease: congestive heart failure > class II New York Heart Association (NYHA); patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Symptomatic or uncontrolled brain metastasis; patients with neurological symptoms must undergo a computed tomography (CT) scan/magnetic resonance imaging (MRI) of the brain to exclude brain metastasis; previously treated brain metastases will be allowed as long as the patient is neurologically stable and is off steroids and anticonvulsants
* Prior radiation to greater than 25% of the bone marrow or whole pelvis radiation
* Patients requiring full therapeutic anticoagulation with warfarin are ineligible because therapy on this trial may result in frequent and recurrent thrombocytopenia; full therapeutic anticoagulation with heparin, low molecular weight heparin, or direct factor Xa inhibitor is permitted
* Patients with a diagnosis of active human immunodeficiency virus (HIV) infection, on anti-retroviral therapy, or with a cluster of differentiation (CD) 4 count less than 200 are ineligible; testing is not required in the absence of clinical findings or suspicion
* Patients with a diagnosis of chronic hepatitis B are ineligible
* Active clinically serious infection > Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or systemic infection requiring IV antibiotic therapy within 14 days preceding the first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first dose of study drug
* Known or suspected allergy to gemcitabine or MLN8237, or any agent given in the course of this trial
* Any clinically significant medical or psychiatric condition that would interfere with protocol treatment
* Prior allogeneic bone marrow or organ transplantation
* Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen
* Requirement for constant administration of proton pump inhibitor or H2 antagonist; intermittent uses of antacids or H2 antagonists are allowed
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Female subject is pregnant or breast-feeding; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patient has received other investigational drugs with 14 days before enrollment
* Other severe acute or chronic medical or psychiatric condition, including uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, requirement for pancreatic enzymes, any condition that would modify small bowel absorption of oral medications, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study
* Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of MLN8237 and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-08-09 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) defined as any related (possibly, probably, or definitely) grade 3 non-hematological toxicity or any attributable grade 4 toxicity graded according to the National Cancer Institute (NCI) CTCAE version 4.0 | Up to 21 days

SECONDARY OUTCOMES:
Incidence of adverse events graded according to NCI CTCAE version 4.0 | Up to 30 days after completion of treatment
  Toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by grade and nadir or maximum values for the laboratory measures), time of onset (i.e. course number), duration, and reversibility or outcome. Frequencies will be reported, with exact 95% confidence intervals. Tables will be created to summarize these toxicities and side effects by dose and by course.
Response rate according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 | Assessed up to 2 years
  Survival will be summarized with Kaplan-Meier plots to describe the outcome of patients treated on this protocol. Median survival time will be estimated using standard life table methods.
Progression Free Survival | Assessed up to 2 years
  Summarized with Kaplan-Meier plots. Median survival time will be estimated using standard life table methods.
Maximum-tolerated dose (MTD) defined as the maximum dose level at which less than 2 patients experience DLT graded according to NCI CTCAE version 4.0 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kelly, Principal Investigator — UC Davis Comprehensive Cancer Center
Locations (1):
- UC Davis Comprehensive Cancer Center, Sacramento, California, United States

REFERENCES:
- See also: University of California Davis Comprehensive Cancer Center — http://www.ucdmc.ucdavis.edu/cancer/